CLINICAL TRIAL: NCT00106171
Title: A Randomized Trial of HAART in Acute/Early HIV Infection
Brief Title: Anti-HIV Medications for People Recently Infected With HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01AI056990-01A1 (NIH); 1R01AI056990-01A1 (NIH)
Record Dates: First submitted 2005-03-21; First posted 2005-03-22 (Estimated); Results first posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections
Keywords: HIV; Acute/Early Seroconverters; Acute Infection; Treatment Naive; Primary HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active

ARMS (2):
- Immediate Treatment Arm (Experimental): Participants will receive immediate HAART for 1 year; then HAART will stopped until clinically indicated.
  Interventions: Drug: Highly active antiretroviral therapy (HAART)
- Deferred Treatment Arm (No Intervention): Participants will receive no immediate HAART, but will receive HAART when HAART is clinically indicated.

INTERVENTIONS:
Drug: Highly active antiretroviral therapy (HAART) — Regimens will be assigned by investigators
  Arms: Immediate Treatment Arm

SUMMARY:
It is not known if anti-HIV treatment for recently infected patients improves long-term patient prognosis. The purpose of this study is to determine if a one year course of anti-HIV medications slows progression of HIV disease in adults recently infected with HIV.

Study hypothesis: A one-year course of HAART administered during acute or early seroconversion may slow the progression of HIV infection.

DETAILED DESCRIPTION:
Although some doctors favor starting anti-HIV treatment as soon as possible after patients learn they are infected, it is not known if treatment for recently infected patients results in slower progression of HIV disease. This study will compare the virologic outcomes of recently infected adults who receive highly active antiretroviral therapy (HAART) with those who receive no treatment. This study will also compare the effects of treatment on patients who enroll within 3 months of seroconversion (acute seroconverters) with patients who enroll within 3 to 12 months of seroconversion (early seroconverters).

This study will last at least 3 years. Participants will be randomly assigned to one of two groups. Group 1 will receive HAART for 1 year; Group 2 will receive no treatment. There will be at least 20 study visits over the 3-year study period. Blood collection will occur at all study visits. A physical exam, medical and medication history, and risk behavior assessment will occur at most visits; participants will also be asked to complete an adherence questionnaire at most visits.

ELIGIBILITY:
Inclusion Criteria:

* Documented acute or recent HIV infection (infected in the past 12 months) as defined in the study protocol
* Antiretroviral naive. Participants who have taken antiretrovirals for postexposure prophylaxis are eligible for this study.
* Able to swallow tablets or capsules
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* Physician unable to design a potentially effective HAART regimen based on results of genotypic resistance testing
* Two CD4 counts of less than 350 cells/mm3 obtained at least 7 days apart within 30 days of study entry
* Viral load less than 5,000 copies/ml within 30 days of study entry in participants who have been infected with HIV-1 for more than six months prior to study entry
* Use of systemic cancer chemotherapy, systemic investigational agents, specific antiretroviral medications, or immunomodulators (growth factors, systemic corticosteroids, HIV vaccines, immune globulin, interleukins, interferons) within 30 days prior to study entry
* Current alcohol or drug use that, in the opinion of the investigator, would interfere with the study
* Serious illness requiring systemic treatment or hospitalization until participant either completes therapy or is clinically stable on therapy for at least 7 days prior to study entry
* Currently involuntarily incarcerated for treatment of either a psychiatric or physical (e.g., infectious disease) illness
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2005-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph B. Margolick, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (5):
- Johns Hopkins University, Baltimore, Maryland, United States
- Canada (4):
  - University of British Columbia, Vancouver, British Columbia
  - Sunnybrook Health Sciences Ctr., Toronto, Ontario
  - Canadian Immunodeficiency Research Collaborative (CIRC) Inc., Toronto, Ontario
  - CHUM - Hotel-Dieu, Montreal, Quebec

REFERENCES:
- [Result] Margolick JB, Apuzzo L, Singer J, Wong H, Lee T, Gallant JE, El-Helou P, Loutfy MR, Rachlis A, Fraser C, Kasper K, Tremblay C, Tossonian H, Conway B. A Randomized Trial of Time-Limited Antiretroviral Therapy in Acute/Early HIV Infection. PLoS One. 2015 Nov 24;10(11):e0143259. doi: 10.1371/journal.pone.0143259. eCollection 2015. PMID 26600459

RESULTS

PARTICIPANT FLOW:
Groups:
- Treated Arm: Participants will receive HAART for 1 year
  Highly active antiretroviral therapy (HAART): Regimens will be assigned by investigators
- Untreated Arm: Participants will receive no treatment
Period: Overall Study
Arm/Group | Treated Arm | Untreated Arm
Started | 57 | 56
Completed | 37 | 46
Not Completed | 20 | 10

BASELINE CHARACTERISTICS:
Groups:
- Immediate Treatment Arm: Participants will receive HAART for 1 year
  Highly active antiretroviral therapy (HAART): Regimens will be assigned by investigators
- Deferred Treatment Arm: Participants will receive no treatment
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment Arm | Deferred Treatment Arm | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.7 [26.1 to 42.3] | 32.8 [27.2 to 44.4] | 33.2 [26.7 to 43.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 52 | 47 | 99
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 27 | 30 | 57
  United States | 30 | 26 | 56

OUTCOME MEASURES:

1. Primary Outcome: Total Treatment-free Time to Initiation of Permanent HAART
Description: All HAART-free time from initial infection with HIV to initiation of permanent HAART
Time Frame: Through study completion, an average of 18 months
Measure: Mean (Full Range); unit: months
Arm/Group | Immediate Treatment Arm | Deferred Treatment Arm
Number analyzed (Participants) | 57 | 56
months | 18 [2 to 22] | 18 [1 to 34]

2. Secondary Outcome: Toxicity as Assessed by the of Number of Participants With Serious Adverse Events
Description: Number of participants with serious adverse events (grade 3 or 4 as defined by the NIH toxicity scale)
Time Frame: Throughout study completion, an average of 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Treatment Arm | Deferred Treatment Arm
Number analyzed (Participants) | 57 | 56
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: through study completion, an average of 18 months
Arm/Group | Immediate Treatment Arm | Deferred Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/56
Other Adverse Events (participants affected / at risk) | 0/57 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No